CLINICAL TRIAL: NCT06670313
Title: Effects of Preoperative and Postoperative Errector Spinal Plan (ESP) Block on Postoperative Analgesia Score, Hemodynamic Response and Patient Satisfaction in Patients Undergoing Laparoscopic Cholecystectomy Surgery
Brief Title: Effect of Preop and Postop ESP Block on Analgesia, Hemodynamics and Patient Satisfaction in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veli Fahri Pehlivan, Assistant Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sait
Record Dates: First submitted 2024-10-25; First posted 2024-11-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Erector Spinae Plane Block

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind: Participants were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preop Erector spinae plane block (Active Comparator): Patients who underwent erector spinae block before surgery
  Interventions: Other: postop Erector spinae plane block
- postop Erector spinae plane block (Active Comparator): Patients who underwent erector spinae block without waking the patient at the end of surgery
  Interventions: Other: postop Erector spinae plane block

INTERVENTIONS:
Other: postop Erector spinae plane block — Postoperative ESP block was performed as the control group

SUMMARY:
Erector spinae plane (ESP) block is an interfascial plane block applied to the paraspinal region, which provides effective visceral and extensive somatic analgesia by providing paravertebral spread of the administered local anesthetic to three and four vertebral levels cranial and caudal. ESP block is a new regional anesthesia method applied with ultrasound (USG) guidance to provide analgesia for various surgeries and for acute or chronic pain. The application of this block is simple and can be performed in the preoperative waiting area with light sedation or no sedation. ESP block can be applied with a single injection or as a continuous infusion by catheter placement.

DETAILED DESCRIPTION:
Erector spinae plane (ESP) block is an interfascial plane block applied to the paraspinal region, which provides effective visceral and extensive somatic analgesia by providing paravertebral spread of the administered local anesthetic to three and four vertebral levels cranial and caudal. ESP block is a new regional anesthesia method applied with ultrasound (USG) guidance to provide analgesia for various surgeries and for acute or chronic pain. The application of this block is simple and can be performed in the preoperative waiting area with light sedation or no sedation. ESP block can be applied with a single injection or as a continuous infusion by catheter placement. The first report related to this block was published in 2016; the block was performed to reduce thoracic neuropathic pain in a patient with metastatic rib disease and rib fracture. So far, the block has been reported to be performed successfully in many cases, including the Nuss procedure, thoracotomies, percutaneous nephrolithotomies, ventral hernia surgeries, and even lumbar fusions.

ELIGIBILITY:
Inclusion Criteria:

* According to the physical classification of the American Society of Anesthesiologists (ASA), ASA I-II group,
* between the ages of 18-65,

Exclusion Criteria:

* Patients who do not want to participate in the study;
* BMI >30,
* Patients with contraindications for ESP block,
* Uncooperative patients,
* Those with renal failure,
* Those with hepatic failure and
* ASA III-IV-V group patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
primary outcome | one day
  1. Systolic arterial pressure,

SECONDARY OUTCOMES:
Sevondary outcome | one day
  1. Postoperative NRS (Numerical pain scale) score,

CONTACTS AND LOCATIONS:
Locations (1):
- Veli Fahri Pehlivan, Sanliurfa, Turkey (Türkiye)